CLINICAL TRIAL: NCT03974802
Title: Refitting Somofilcon A Sphere Contact Lens Wearers Into Fanfilcon A Sphere Lenses for 4-Weeks of Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EX-MKTG-101
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: First pair of study lenses (habitual lenses) will be dispensed and worn for 4 weeks for daily wear, then second pair of lenses (test lenses) will be dispensed and worn for 4 weeks for daily wear.
Masking Description: Study lenses will be transferred, by an assistant, out of their packaging to unmarked new contact lens cases filled with unpreserved sterile saline just prior to dispensing to maintain subject masking of the study lenses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- somofilcon A (habitual) lens, then fanfilcon A (test) lens (Experimental): Participants are habitual wearers of somofilcon A lens and refitted with fanfilcon A lens.
  Interventions: Device: somofilcon A contact lens; Device: fanfilcon A contact lens

INTERVENTIONS:
Device: somofilcon A contact lens — Contact Lens
  Other Names: clariti elite; Habitual lens
Device: fanfilcon A contact lens — Contact Lens
  Other Names: Avaira Vitality; Test lens

SUMMARY:
The aim of this subject-masked prospective study is to evaluate the clinical performance of habitual wearers of Clariti Elite sphere lenses after a refit with Avaira Vitality sphere lenses.

DETAILED DESCRIPTION:
The aim of this subject-masked prospective study is to evaluate the clinical performance of habitual wearers of Clariti Elite sphere lenses after a refit with Avaira Vitality sphere lenses for 4 weeks of daily wear.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft contact lens wearer
* Has a contact lens spherical prescription between - 0.25 to - 8.00 (inclusive)
* Have no less than -0.75D of astigmatism in both eyes.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Patient contact lens refraction should fit within the available parameters of the study lenses.
* Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Has a CL prescription outside the range of the available parameters of the study lenses.
* Has a spectacle cylinder of ≥ 1.00D in either eye.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
* Presence of clinically significant (grade 2-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (past or present)
  * Seborrheic eczema, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Velázquez Guerrero, MSc., FIACLE, Principal Investigator — School of Optometry, National Autonomous University (UNAM), Mexico City
Locations (1):
- Optometry Clinic, National Autonomous University, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Somofilcon A (Habitual) Lens, Then Fanfilcon A (Test) Lens: Participants wore somofilcon A lens (habitual) for 4- weeks and refitted with fanfilcon A lens (test) for 4-weeks.
  somofilcon A contact lens: Contact Lens
  fanfilcon A contact lens: Contact Lens
Period: Overall Study
Arm/Group | Somofilcon A (Habitual) Lens, Then Fanfilcon A (Test) Lens
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Participants wore somofilcon A lens (habitual) for 4- weeks and refitted with fanfilcon A lens (test) for 4-weeks.
  somofilcon A contact lens: Contact Lens
  fanfilcon A contact lens: Contact Lens
Arm/Group | Overall Study
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 41

OUTCOME MEASURES:

1. Primary Outcome: Lens Centration for Somofilcon A (Habitual) Lens
Description: Lens Centration was measured using a 3-point scale (1=optimal centration, 2=decentration acceptable, 3=decentration unacceptable).
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Groups:
- Somofilcon A (Habitual) Lens: Participants wore their habitual somofilcon A lens for 4-weeks.
  somofilcon A: Contact lens
Arm/Group | Somofilcon A (Habitual) Lens
Number analyzed (Participants) | 41
percentage of participants
  Optimum | 100
  Decentration Acceptable | 0
  Decentration Unacceptable | 0

2. Primary Outcome: Lens Centration for Somofilcon A (Habitual) Lens
Description: as for outcome 1
Time Frame: 4- weeks
Measure: Number; unit: percentage of participants
Arm/Group | Somofilcon A (Habitual) Lens
Number analyzed (Participants) | 41
percentage of participants
  Optimum | 100
  Decentartion Acceptable | 0
  Decentration Unacceptable | 0

3. Primary Outcome: Lens Centration for Fanfilcon A (Test) Lens
Description: as for outcome 1
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Groups:
- Fanfilcon A (Test) Lens: Participants were refitted with fanfilcon A test lens for 4-weeks.
  fanfilcon A: Contact lens
Arm/Group | Fanfilcon A (Test) Lens
Number analyzed (Participants) | 41
percentage of participants
  Optimum | 100
  Decentration Acceptable | 0
  Decentration Unacceptable | 0

4. Primary Outcome: Lens Centration for Fanfilcon A (Test) Lens
Description: as for outcome 1
Time Frame: 2-weeks
Measure: Number; unit: percentage of participants
Arm/Group | Fanfilcon A (Test) Lens
Number analyzed (Participants) | 41
percentage of participants
  Optimum | 100
  Decentration Acceptable | 0
  Decentration Unacceptable | 0

5. Primary Outcome: Lens Centration for Fanfilcon A (Test) Lens
Description: Lens Centration was measured using a 3-point scale(1=optimal centration, 2=decentration acceptable, 3=decentration unacceptable).
Time Frame: 4- weeks
Measure: Number; unit: percentage of participants
Arm/Group | Fanfilcon A (Test) Lens
Number analyzed (Participants) | 41
percentage of participants
  Optimum | 100
  Decentration Acceptable | 0
  Decentration Unacceptable | 0

6. Primary Outcome: Lens Corneal Coverage for Somofilcon A (Habitual) Lens
Description: Lens Corneal Coverage was rated as either Yes or No (Yes = full corneal coverage all time / no= incomplete corneal coverage)
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Somofilcon A (Habitual) Lens
Number analyzed (Participants) | 41
percentage of participants
  Yes | 100
  No | 0

7. Primary Outcome: Lens Corneal Coverage for Somofilcon A (Habitual) Lens
Description: as for outcome 6
Time Frame: 4 -weeks
Measure: Number; unit: percentage of participants
Arm/Group | Somofilcon A (Habitual) Lens
Number analyzed (Participants) | 41
percentage of participants
  Yes | 100
  No | 0

8. Primary Outcome: Lens Corneal Coverage for Fanfilcon A (Test) Lens
Description: as for outcome 6
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Groups:
- Fanfilcon A (Test) Lens: Participants were refitted with fanfilcon A lens (test) for 4-weeks.
  fanfilcon A: Contact lens
Arm/Group | Fanfilcon A (Test) Lens
Number analyzed (Participants) | 41
percentage of participants
  Yes | 100
  No | 0

9. Primary Outcome: Lens Corneal Coverage for Fanfilcon A (Test) Lens
Description: as for outcome 6
Time Frame: 2-weeks
Measure: Number; unit: percentage of participants
Arm/Group | Fanfilcon A (Test) Lens
Number analyzed (Participants) | 41
percentage of participants
  Yes | 100
  No | 0

10. Primary Outcome: Lens Corneal Coverage for Fanfilcon A (Test) Lens
Description: as for outcome 6
Time Frame: 4-weeks
Measure: Number; unit: percentage of participants
Arm/Group | Fanfilcon A (Test) Lens
Number analyzed (Participants) | 41
percentage of participants
  Yes | 100
  No | 0

11. Primary Outcome: Percentage of Lens Tightness for Somofilcon A (Habitual) Lens
Description: Lens Tightness: Push Up Test measured by 0% to 100% continuous scale (0%-falls from cornea without lid support, 50% = optimum, and 100% = no movement)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A (Habitual) Lens
Number analyzed (Participants) | 41
units on a scale | 51.7 (5.0)

12. Primary Outcome: Percentage of Lens Tightness for Somofilcon A (Habitual) Lens
Description: as for outcome 11
Time Frame: 4-Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A (Habitual) Lens
Number analyzed (Participants) | 41
units on a scale | 51.8 (5.0)

13. Primary Outcome: Percentage of Lens Tightness for Fanfilcon A (Test) Lens
Description: as for outcome 11
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fanfilcon A Lens (Test): Participants were refitted with fanfilcon A lens (test) for 4-weeks.
  fanfilcon A: Contact lens
Arm/Group | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 41
units on a scale | 50.5 (2.2)

14. Primary Outcome: Percentage of Lens Tightness for Fanfilcon A (Test) Lens
Description: as for outcome 11
Time Frame: 2-Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 41
units on a scale | 50.4 (1.7)

15. Primary Outcome: Percentage of Lens Tightness for Fanfilcon A (Test) Lens
Description: as for outcome 11
Time Frame: 4-Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 41
units on a scale | 50.2 (1.6)

16. Primary Outcome: Post-Blink Movement for Somofilcon A (Habitual) Lens
Description: Post-Blink movement was measured on a scale 0-4 (0=Insufficient, unacceptable movement, 4 = Excessive, unacceptable movement)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A (Habitual) Lens
Number analyzed (Participants) | 41
units on a scale | 1.95 (0.2)

17. Primary Outcome: Post-Blink Movement for Somofilcon A (Habitual) Lens
Description: as for outcome 16
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A (Habitual) Lens
Number analyzed (Participants) | 41
units on a scale | 1.95 (0.2)

18. Primary Outcome: Post-Blink Movement for Fanfilcon A (Test) Lens
Description: as for outcome 16
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 41
units on a scale | 1.95 (0.2)

19. Primary Outcome: Post-Blink Movement for Fanfilcon A (Test) Lens
Description: as for outcome 16
Time Frame: 2-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 41
units on a scale | 2.00 (0.0)

20. Primary Outcome: Post-Blink Movement for Fanfilcon A (Test) Lens
Description: as for outcome 16
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 41
units on a scale | 2.00 (0.0)

21. Primary Outcome: Overall Lens Fit Acceptance for Somofilcon A (Habitual) Lens
Description: Overall fit acceptance was measured using a scale of 0-4 (0= should not be worn, 1 = borderline but unacceptable, 2 = min. acceptable, early review, 3 = not perfect but OK to dispense, and 4 = perfect)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A (Habitual) Lens
Number analyzed (Participants) | 41
units on a scale | 3.85 (0.4)

22. Primary Outcome: Overall Lens Fit Acceptance for Somofilcon A (Habitual) Lens
Description: as for outcome 21
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A (Habitual) Lens
Number analyzed (Participants) | 41
units on a scale | 3.83 (0.5)

23. Primary Outcome: Overall Lens Fit Acceptance for Fanfilcon A (Test) Lens
Description: as for outcome 21
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 41
units on a scale | 3.95 (0.2)

24. Primary Outcome: Overall Lens Fit Acceptance for Fanfilcon A (Test) Lens
Description: as for outcome 21
Time Frame: 2-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 41
units on a scale | 3.98 (0.2)

25. Primary Outcome: Overall Lens Fit Acceptance for Fanfilcon A (Test) Lens
Description: as for outcome 21
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 41
units on a scale | 3.98 (0.2)

26. Secondary Outcome: Average Daily Wearing Time - Somofilcon A (Habitual) Lens
Description: Average Daily Wearing Time for somofilcon A (Habitual) lens - measured by time hours/day
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Somofilcon A (Habitual) Lens
Number analyzed (Participants) | 41
hours/day | 12.1 (3.1)

27. Secondary Outcome: Average Daily Wearing Time - Fanfilcon A (Test) Lens
Description: Average daily wearing time for fanfilcon A (test) lens was measured in hours/day
Time Frame: 2-weeks
Measure: Mean (Standard Deviation); unit: hours/day
Groups:
- Fanfilcon A Lens (Test): Participants were refitted with Participants were refitted with fanfilcon A lens (test) for 4-weeks.
  fanfilcon A: Contact lens
Arm/Group | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 41
hours/day | 12.3 (2.0)

28. Secondary Outcome: Average Daily Wearing Time - Fanfilcon A (Test) Lens
Description: Average daily wearing time for fanfilcon A (test) lens was measured in hours/day
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 41
hours/day | 12.3 (2.0)

29. Secondary Outcome: Average Comfortable Wearing Time - Somofilcon A (Habitual) Lens
Description: Average Comfortable Wearing Time - somofilcon A (habitual) Lens measured in hours/day. Assessed using typical time of day when subject first experiences lens awareness or irritation.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Somofilcon A (Habitual) Lens
Number analyzed (Participants) | 41
hours/day | 9.8 (3.3)

30. Secondary Outcome: Average Comfortable Wearing Time - Fanfilcon A (Test) Lens
Description: Average Comfortable Wearing Time - fanfilcon A (test) Lens measured in hours/day. Assessed using typical time of day when subject first experiences lens awareness or irritation.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 41
hours/day | 10.6 (2.2)

31. Secondary Outcome: Average Comfortable Wearing Time - Fanfilcon A (Test) Lens
Description: as for outcome 30
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 41
hours/day | 10.8 (1.8)

ADVERSE EVENTS:
Time Frame: From dispense up to 4-weeks for each study lens
Groups:
- Somofilcon A (Habitual) Lens: Subjects wore their habitual somofilcon A lens for 4 -weeks.
  somofilcon A contact lens: Contact Lens
- Fanfilcon A (Test) Lens: Subjects were refitted with fanfilcon A lens (test) for 4- weeks.
  fanfilcon A contact lens: Contact Lens
Arm/Group | Somofilcon A (Habitual) Lens | Fanfilcon A (Test) Lens
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT03974802/Prot_SAP_000.pdf